CLINICAL TRIAL: NCT04535479
Title: Neurophysiological Characterization of Dry Needling in People With Spasticity Due to Stroke
Brief Title: Dry Needling for Spasticity in Stroke
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Aiko Thompson, Associate Professor, Medical University of South Carolina
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00095077-A
Record Dates: First submitted 2020-08-27; First posted 2020-09-02 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Stroke; Muscle Spasticity
Keywords: Dry Needling; Nervous System; Central Nervous System
MeSH Terms: conditions — Stroke; Muscle Spasticity; Neurologic Manifestations | interventions — Dry Needling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Individuals with spasticity resulting from stroke (Experimental): This is an experimental intervention in which individuals will receive dry needling to relieve spasticity in the target muscle. The study team will examine the effects of this treatment on the nervous system by performing assessments just prior to, immediately after, 90 minutes after, and 72 hours after dry needling. These assessments will examine how you move your arm or leg and how your nervous system responds to non-invasive nerve stimulation.
  Interventions: Behavioral: Dry Needling
- Individuals with no known neurological injury (Experimental): This is an experimental intervention in which individuals will receive dry needling of an arm or leg muscle. The study team will examine the effects of this treatment on the nervous system by performing assessments just prior to, immediately after, 90 minutes after, and 72 hours after dry needling. These assessments will examine how you move your arm or leg and how your nervous system responds to non-invasive nerve stimulation.
  Interventions: Behavioral: Dry Needling

INTERVENTIONS:
Behavioral: Dry Needling — Dry needling is a procedure in which a thin, stainless steel needle is inserted into the skin to produce a muscle twitch response. It is intended to release a knot in a muscle and relieve pain.

SUMMARY:
The study team is recruiting 20 adults with spasticity due to chronic stroke and 20 adults with no neurological injuries for a 2 day study. In people with chronic stroke, one of the most common and disabling problems is spasticity (increased muscle tone or muscle stiffness). The purpose of this research study is to examine effects of dry needling on the nervous system (pathways between the muscle, spinal cord, and brain) in people with spasticity due to chronic stroke. Dry needling is a procedure in which a thin, stainless steel needle is inserted into your skin to produce a muscle twitch response. It is intended to release a knot in your muscle and relieve pain.

The total study duration is 2 days. The first visit will take about 3 hours, during which dry needling will take place, and the second visit will take about 1 hour. During both visits you will be asked to participate in examinations of reflexes (muscle responses to non-invasive nerve stimulation) and arm/leg function.

ELIGIBILITY:
Inclusion Criteria:

For adults with no known neurological conditions:

* ≥18 years old
* no known neurological injuries.

For individuals after stroke:

* neurologically stable for >6 months (and >1 yr post stroke)
* medical clearance to participate
* unilateral ankle and/or wrist spasticity, confirmed by Modified Ashworth Scale (MAS) > 1 and the presence of spastic hyperreflexia

Exclusion Criteria:

* motoneuron injury (i.e. the neurons that give rise to the axons innervating the muscles) with inadequate response to stimulation
* a cardiac condition ( history of myocardial infarction, congestive heart failure, pacemaker use, coronary artery disease, atrial fibrillation, congenital heart disease, uncontrolled hypertension)
* a medically unstable condition (including temporary infections and pregnancy)
* age <18 years old
* cognitive impairment sufficient to interfere with informed consent or successful completion of the protocol
* metal allergies
* needle phobias
* lymphedema over a limb (due to risk of infection/cellulitis)
* abnormal bleeding tendencies
* compromised immune system
* vascular disease
* uncontrolled diabetes
* history of epilepsy (as DDN generates strong somatosensory sensation)
* anxiety disorders or in distress.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in the H-reflex amplitude in response to nerve stimulation | baseline, immediately after DDN, 90 minutes after DDN, and 72 hours after DDN
  H-reflex amplitude (mV) reflects the excitability of its reflex pathway. Changes in the H-reflex amplitude indicate that DDN influences the spinal reflex excitability. In the lower extremity this will be measured in the tibialis anterior and the triceps surae. In the upper extremity this will be measured in flexor carpi ulnaris and flexor carpi radialis.
2. Changes in cutaneous reflexes elicited by non-noxious stimulation of cutaneous or mix nerves | baseline, immediately after DDN, 90 minutes after DDN, and 72 hours after DDN
  Changes in the cutaneous reflex amplitudes would indicate that DDN can influence the spinal processing of cutaneous information.
3. Changes in perception of cutaneous stimuli as measured by perception and radiating threshold of cutaneous nerve stimulation | baseline, immediately after DDN, 90 minutes after DDN, and 72 hours after DDN
  Changes in thresholds of cutaneous nerve stimulation would imply that DDN can affect the perception of cutaneous input.

SECONDARY OUTCOMES:
Change in ability to move the arm or leg as measured by the Fugl-Meyer Assessment (FMA) | baseline, 90 minutes after DDN, and 72 hours after DDN
  An increase in the FMA score indicates better movement of the arm or leg.
Change in spasticity as measured by the Modified Ashworth Scale (mAS) | baseline, 90 minutes after DDN, and 72 hours after DDN
  The mAS score ranges from 0: normal muscle tone to 4: rigid in flexion or extension. A decrease in mAS indicates decreased spasticity.
Change in the ability to move the limb as measured by range of motion (ROM) | baseline, immediately after DDN, 90 minutes after DDN, and 72 hours after DDN
  ROM is measured in degrees using a standard goniometer. Increased ROM, which will be measured both passively (moved by the assessor) and actively (participant moves the arm themselves), indicates improved ability to move the limb.
Change in pain level as measured by the visual analog scale (VAS) for pain | baseline, immediately after DDN, 90 minutes after DDN, and 72 hours after DDN
  Pain is rated by the participant on a scale from 0 (no pain) to 10 (worst pain imaginable). Decreased score on the VAS for pain indicates decreased pain.

CONTACTS AND LOCATIONS:
Overall Officials: Aiko K Thompson, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No